CLINICAL TRIAL: NCT06310330
Title: Technology Revising Ultrasound Solutions for Tomorrow - Anticancer-treatment Cardiotoxicity Identification by Echocardiography
Brief Title: TRUST-ACE - Anticancer-treatment Cardiotoxicity Identification by Echocardiography
Acronym: TRUST-ACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/1059
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Breast Neoplasm Malignant Primary
Keywords: echocardiography; breast cancer; artificial intelligence; cardiotoxicity
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Intervention Model Description: Randomization 1:1 to two different modes of follow-up
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Standard of care echocardiographic follow-up
  Interventions: Diagnostic Test: Comprehensive echocardiographic follow-up
- Simplified care (Experimental): Simplified echocardiographic follow-up
  Interventions: Diagnostic Test: Simplified echocardiographic follow-up

INTERVENTIONS:
Diagnostic Test: Comprehensive echocardiographic follow-up — Comprehensive echocardiographic follow-up for identification of CRTCD in breast cancer patients
  Arms: Usual care
Diagnostic Test: Simplified echocardiographic follow-up — Simplified echocardiographic follow-up for identification of CRTCD in breast cancer patients
  Arms: Simplified care

SUMMARY:
TRUST-ACE will compare a simplified echocardiographic protocol focusing on ventricular function with the guideline recommended comprehensive echocardiographic examination using a randomised design in follow-up of breast-cancer patients with respect to identification of cancer treatment related cardiac dysfunction (CTRCD).

Secondly, the study will evaluate whether novel tools used to improve standardization of recordings as well as automated measurements of central measurements, e.g. ejection fraction (EF) and global longitudinal strain (GLS) can improve the precision of echocardiography in daily clinical practice.

DETAILED DESCRIPTION:
Cancer treatment related cardiac dysfunction (CTRCD) is a well-known complication to cancer treatment with implication both with respect to treatment and prognosis of the cancer as well as heart.

CTRCD, often named cardiotoxicity, usually refers to myocardial dysfunction and heart failure developing after administration of potentially cardiotoxic therapy. By precise diagnostics, adequate treatment can be started early to prevent heart failure and unnecessary discontinuation of the potential life-saving cancer treatment may be avoided. However, guideline advocated analyses of cardiac function (EF and GLS) by echocardiography are time consuming and many operators base their semi-quantitative estimates on visual assessment. Furthermore, test-retest variability for both EF and GLS are significant and may exceed the guideline recommended cut-offs for identification of cancer therapy-related cardiovascular toxicity.

The study will compare a simplified echocardiographic protocol focusing on ventricular function with the guideline recommended comprehensive echocardiographic examination using a randomized design. The study will also evaluate if novel tools for improved standardization of recordings and automated measurements of relevant measurements as ejection fraction (EF) and global longitudinal strain (GLS) can improve the diagnostic precision.

Breast cancer patients referred for follow-up at the echocardiography will be included.

Patients will be randomized 1:1 to A) examinations with two- and three-dimensional echocardiography including all central measures of cardiac size and function measured by sonographers as recommended by the European guidelines and as clinical practice or B) echocardiographic examinations focusing on the ventricles.

Subpopulations will undergo additional testing with serial echocardiographic examinations by four operators on the same day with and without use of novel tools for improved standardization of recordings and automated measurements.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer and referral for follow-up to identify potential CTRCD

Exclusion Criteria:

* Not willing or able to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients correctly classified with cancer therapy related cardiac dysfunction (CTRCD) | 15 months
  Cancer treatment related cardiac dysfunction

OTHER OUTCOMES:
Proportion of patients misclassified as having/not having cancer therapy related cardiac dysfunction (CTRCD) | 15 months
  Proportion of misclassified CTRCD
Risk classification | 0 days
  Risk classification for identification of CTRCD
Risk classification | 15 months
  Risk classification for identification of CTRCD
Test-retest variability, systolic left ventricular size and function | 0 days
  Test-retest variability of systolic left ventricular size and function
Test-retest variability, systolic left ventricular size and function | 15 months
  Test-retest variability systolic left ventricular size and function
Test-retest variability, diastolic left ventricular size and function | 0 days
  Test-retest variability of diastolic left ventricular function
Test-retest variability, diastolic left ventricular size and function | 15 months
  Test-retest variability of diastolic left ventricular size and function
Test-retest variability, right ventricular size and function | 0 days
  Test-retest variability of right ventricular size and function
Test-retest variability, right ventricular size and function | 15 months
  Test-retest variability of right ventricular size and function
Time consumption | 0 days
  Time used for echocardiographic examination
Time consumption | 15 days
  Time used for echocardiographic examination

CONTACTS AND LOCATIONS:
Overall Officials: Espen Holte, MD, PhD, Principal Investigator — St. Olavs Hospital
Locations (1):
- St. Olavs hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sabo S, Pettersen H, Boen GC, Jakobsen EO, Langoy PK, Nilsen HO, Pasdeloup D, Smistad E, Ostvik A, Lovstakken L, Stolen S, Grenne B, Dalen H, Holte E. Real-time guidance and automated measurements using deep learning to improve echocardiographic assessment of left ventricular size and function. Eur Heart J Imaging Methods Pract. 2025 Jul 21;3(2):qyaf094. doi: 10.1093/ehjimp/qyaf094. eCollection 2025 Jul. PMID 40747448